CLINICAL TRIAL: NCT07107594
Title: Multimodal Intervention During Neoadjuvant Chemotherapy in Patients With Early-breast Cancer as a Strategy to Improve Treatment Response: DIANA Trial (Multimodal Prehabilitation: DIet, ANxiety Control Psychotherapy, Physical Activity)
Brief Title: Multimodal Prehabilitation Program That Combines Physical Exercise, Psychological Intervention and Nutritional Support to Improve the Response to Neoadjuvant Chemoterhapy in Early Breast Cancer Patients
Acronym: DIANA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Helena Castillo, Medical Doctor (MD), Specialized in Gynecology and Obstetrics, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2023/1036
Record Dates: First submitted 2025-07-06; First posted 2025-08-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Prehabilitation
Keywords: Breast cancer; Early breast cancer; Prehabilitation; Multimodal prehabilitation; Neoadjuvant chemotherapy; Lifestyle; Quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The pathologist responsible for analyzing the pathological response to the treatment will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 107 women that will follow the standard of care. Patients in the control group will receive proper information and recommendations about lifestyle modifications according to the most recent oncological guidelines. The benefits of physical exercise, a healthy diet and psychological support will be exposed, but such interventions will not be provided in our centre.
- Prehabilitation (Experimental): 107 women that will follow the multimodal prehabilitation program during NACT (physical exercise, psychological intervention, nutritional support).
  Interventions: Behavioral: Multimodal prehabilitation

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — Multimodal prehabilitation program during NACT (4-6 months) that will combine: 1) Physical exercise: cardiovascular and strength exercises designed by specialized physiotherapists, structured in 1-hour sessions twice a week. The characteristics of the activity will be adapted to the treatment phase and the physical condition of each woman. 2) Psychological therapies: standardized mindfullness practice by a specialized psychologist. As an alternative, patients who refuse mindfullness could receive psychological sessions on stress and anxiety management. 3) Nutritional counseling: periodic sessions with a specialized nutritionist providing dietary recommendations and nutritional advice adapted to the disease and condition of the patients.
  Arms: Prehabilitation

SUMMARY:
The aim of this clinical trial is to evaluate whether following a multimodal prehabilitation program including physical exercise, nutritional support and psychological intervention during neoadjuvant chemotherapy in breast cancer patients could improve the pathological response to chemotherapy.

214 women with non-metastatic breast cancer with indication of chemotherapy before surgery will be eligible to participate. Patients will be randomly assigned to either the intervention group or the control group.

* Patients assigned to the intervention group (107 women) will undergo a directed multimodal prehabilitation program during the chemotherapy (4-6 months), including structured physical exercise, psychological intervention and nutritional guidance.
* Patients assigned to the control group (107 women) will undergo standard clinical management for their disease without multimodal prehabilitation.

The response to chemotherapy between the two groups will be evaluated and compared. It is expected that multimodal prehabilitation will increase the response to chemotherapy and will improve the postoperative recovery of patients and their quality of life, as well as reducing the number of complications from surgery and chemotherapy treatment. Changes in the tumor microenvironment are also expected after prehabilitation.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common neoplasm worldwide and the leading cause of death among women. Neoadjuvant chemotherapy (NACT) is currently one of the main therapeutic pillars. The pathological response after NACT has demonstrated prognostic value in BC, being also a determinant factor for posterior treatments. In recent years, research has increasingly focused on the impact of lifestyle changes on BC, such as physical exercise, diet, and psychological interventions. These actions are part of what is known as prehabilitation, defined as the set of strategies applied prior to surgery to optimize the physical and emotional condition of patients before the surgical intervention.

The individual application of these strategies in BC patients has shown improved oncological outcomes, with positive effects on quality of life and tolerance to medical treatments. Furthermore, evidence suggests that these interventions may favorably modulate the tumor microenvironment by reducing intratumoral hypoxia, enhancing antitumor immune responses, and modulating systemic pro-inflammatory states.

Despite the demonstrated benefits of prehabilitation in multiple medical and surgical fields, there is limited evidence regarding its impact on systemic treatment outcomes in BC patients. There is also a lack of solid evidence evaluating the role of multimodal prehabilitation (combining different prehabilitation strategies) in BC, as well as its effect on treatment response and tolerance.

The current study proposes the application of a multimodal prehabilitation program during the NACT window, based on structured physical exercise, psychological therapy (mindfulness or anxiety-control techniques), and nutritional counseling in BC patients, as a strategy to enhance treatment response through changes in the tumor microenvironment. Additionally, it will be assessed whether the intervention improves treatment tolerance and postoperative recovery, among others.

The study consists of a randomized, single-blind, controlled clinical trial with two parallel groups that will include 214 women diagnosed with non-metastatic breast cancer, eligible for NACT, and awaiting surgery at our center.

Participants will be randomized into two parallel groups in a 1:1 ratio (control and intervention group, including 107 women each). A basal evaluation will be performed in all patients before starting NACT, reporting their physical, nutritional and psychological status, as well as a tumor microenvironment study in the diagnostic biopsy sample. All patients will undergo 4-6 months of NACT, the control group with standard clinical management and the intervention group following the multimodal prehabilitation program. After NACT, the physical, nutritional and psychological status of all patients will be re-evaluated. Patients will undergo surgery according to their disease and the pathological response to the treatment will be assessed.

The primary outcome will be the pathological response after NACT in both groups, assessed through the Residual Cancer Burden (RCB) index. Secondary outcomes will include NACT tolerance, quality of life, psychological and nutritional status, postoperative recovery, tumor microenvironment changes and patients' physical condition.

The group of BC patients undergoing the multimodal prehabilitation program during NACT is expected to achieve better response rates (RCB 0 and I) than the control group. Furthermore, the multimodal intervention is anticipated to promote quantitative and/or qualitative changes in the tumor microenvironment, improve NACT tolerance, enhance quality of life, and optimize postoperative recovery and the patients' physical, psychological, and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-metastatic breast cancer: stages cT1-T4, cN0-N3, M0, and candidates for neoadjuvant chemotherapy (NAC).
* Age ≥ 18 years.
* Signed informed consent.

Exclusion Criteria:

* Contraindication or physical inability to perform moderate-to-high intensity physical exercise.
* Pregnant or breastfeeding patients.
* Presence of other active synchronous neoplasms.
* Metastatic breast cancer (stage IV).
* Patients already engaging in regular physical exercise: more than 150 minutes of moderate or intense aerobic exercise per week.
* Male breast cancer patients.
* Personal history of a previous malignancy treated with chemotherapy.
* Severe or poorly controlled psychiatric illness (including uncontrolled active substance abuse).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Residual Cancer Burden Index (RCB) | From enrollment (baseline, day 1) until the end of treatment at 4-6 months (preoperative).
  The main variable of the trial is the RCB index score, obtained from the histological specimen of the oncological surgery performed after NAC. The four levels of response of the RCB index (RCB 0, I, II and III) will be divided into a favorable profile of response (fRCB), that will include cathegories RCB 0 and I, and an unfavorable response profile (uRCB), including RCB II and III.
  It is estimated that the average rate of a favorable RCB (fRCB) score, including RCB 0 and RCB I, will be approximately 40% in the control arm. Parallelly, the expected rates of unfavorable RCB (uRCB) scores, including RCB II and RCB III, are 60%. The objective is to improve the response rates by 20% in the intervention group, with 60% of fRCB scores and 40% of uRCB scores in this group.

SECONDARY OUTCOMES:
Tumor microenvironment (Gene expression analyses) | From enrollment (baseline, day 1) until the end of treatment at 4-6 months (postoperative).
  Formalin fixed-paraffin embedded tumor tissue blocks will be analyzed by hematoxylin and eosin staining, to check tumor surface area. Samples with ≥20% of tumor cells will be selected for RNA extraction. The High Pure FFPET RNA Isolation Kit (Roche) will purify RNA from FFPE tumor samples. A minimum of ∼100 ng of total RNA will be used to measure the expression of 185 breast cancer-related and immune-related genes including the genes of PAM50 and HER2DX and 7 housekeeping genes using the nCounter platform (Nanostring Technologies, Seattle, USA). The gene expression for each sample will be independently normalized to the geometric mean of housekeeping genes. The 14-gene immunoglobulin (IGG) signature (i.e., CD27, CD79A, HLA-C, IGJ, IGKC, IGL, IGLV3-25, IL2RG, CXCL8, LAX1, NTN3, PIM2, POU2AF1 and TNFRSF17) will be calculated.
Tumor staging | At diagnosis or day 1 (clinical TNM or cTNM) and after surgery (pathological TNM or pTNM)
  Registered according to the TNM system by the. American Joint Committee on Cancer (AJCC) 8th edition
Tumor cellularity after NACT | After the surgery (after NACT, 4-6 months from day 1)
  Reported as the percentage (%) of neoplastic cells in the surgical specimen.
Assessment of vascular density in peritumoral areas | At enrollment (baseline, day 1) and at the end of treatment at 4-6 months (postoperative).
  The assessment will involve evaluating microvascular density through immunohistochemical staining for CD31 on tumor or tumor bed sections. This evaluation follows a two-step process:
  1. Hotspot Area Selection: Identification of hotspot areas under a light microscope at 4x magnification.
  2. Manual Counting: Manual counting of all vascular lumens in the selected field at 20x magnification.
  This method ensures precise quantification of vascular density in both the peritumoral and tumor bed regions.
Adverse effects of neoadjuvant chemotherapy | After the treatment (4-6 months later, presurgical).
  They will be recorded by the research team and classified according to the CTCAE (Common Terminology Criteria for Adverse Events) version 5.0. Data will be collected at the end of NAC in both groups.
Chemotherapy completion rate | At the end of the treatment (4-6 months after day 1, preoperative)
  The proportion of patients who received the full course of chemotherapy with the corresponding dose. This will be evaluated before surgery in both groups.
Hospitalization during NACT | At the end of the treatment (4-6 months after day 1, preoperative)
  Need for hospitalization during neoadjuvant chemotherapy: the number of hospital admissions prior to surgery will be recorded as an absolute count.
Post-surgical hospitalization | From the surgery (5-7 months after day 1) until 30 days after the operation.
  Length of hospitalization after oncological surgery: Measured in days.
Pain control after oncological surgery | Since the surgery is done (5-7 months from day 1) until hospital discharge.
  Pain will be assessed using the Visual Analogue Scale (VAS) during the hospital stay. The scale ranges from 0 to 10, with higher scores indicating greater pain severity.
Post-operative complications | From the surgery (5-7 months from day 1) until 30 days after.
  These will be classified based on timing as immediate postoperative complications (during the procedure or within 24 hours), early complications (up to 7 days post-surgery), and late postoperative complications (from 7 to 30 days post-surgery). Severity will be recorded using the Clavien-Dindo scale.
  Emergency visits and readmissions will also be reported: The absolute number, reasons, and length of hospital stay will be recorded up to 30 days post-surgery.
Weight | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), and 1 year after surgery.
  Weight in kilograms will be registered before and after NACT
Body Mass Index | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), and 1 year after surgery.
  Body mass index (BMI) will be measured before and after chemotherapy (kg/m2)
Physical activity level | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical) and 1 year after the surgery.
  The international questionnaire of Physical Activity (IPAQ) will be used to register the level of physical activity of the subjects. Minimum score: 0 MET-min/week. Maximum score: no formal upper limit (normally 20,000 MET-min/week). According to the punctuation, the level of physical activity can be classified into low (< 600 MET-min/week), moderate (≥ 600 and < 3,000 MET-min/week) or high (≥ 3,000 MET-min/week).
Strength | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical) and 1 year after the surgery.
  Assessed through the hand grip strength test, using a hand-held dynamometer (measured in kilograms).
Estimated maximal oxygen uptake (VO2 max) | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical) and 1 year after the surgery.
  To evaluate the general physical status of patients (as an estimate of VO₂), the 30-Second Sit-to-Stand Test will be performed and recorded as an absolute number.
Change in oxygen consumption (VO2) from baseline to post-neoadjuvant therapy | Before the chemotherapy (baseline or day 1) and after the treatment (4-6 months later, presurgical).
  Through a Cardiopulmonary Exercise Testing (CPET), the oxygen consumption will be measured in all patients (ml/kg/min) before and after finishing neoadjuvant chemotherapy.
Patient-perceived quality of life | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), 1 month after surgery and 1 year after the surgery.
  Measured using the EORTC QLQ-30 questionnaire (0-100 points: higher scores on functional scales and the global health status scale indicate better functioning and quality of life, while higher scores on symptom scales indicate a higher level of symptoms).
Anxiety and Depression levels | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), 1 month after surgery and 1 year after the surgery.
  Assessed using the Hospital Anxiety and Depression Scale (HADS), which score ranges from 0 to 21 points. Higher scores indicate more severe symptoms of anxiety or depression: 0-7: Normal or no significant anxiety/depression, 8-10: Mild anxiety/depression, 11-15: Moderate anxiety/depression, 16-21: Severe anxiety/depression.
Mindfulness status | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), and 1 month after surgery.
  Assessed through the Five Facet Mindfulness Questionnaire (FFMQ). Score 39 - 195 points. A higher score indicates a greater level of mindfulness.
Nutritional status | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), and 1 year after the surgery.
  Complete blood analysis: Including liver and renal profile, blood count, ionogram, albumin, prealbumin, glucose, interleukin-6 and IGF-1.
Adherence to mediterranean diet | Before the chemotherapy (baseline or day 1), after the treatment (4-6 months later, presurgical), 1 month after surgery and 1 year after the surgery.
  Validated Questionnaire of Mediterranean Diet Adherence (MEDAS-14). Scoring: 0-14 points. Higher scores mean higher adherence to Mediterranean diet, being a score equal or superior to 9 considered a good adherence to such diet.
Prehabilitation program adherence | After the prehabilitation program (4-6 months from day 1, presurgical).
  Measured by the number of sessions attended relative to the scheduled sessions.
Body image perception | 1 year after the surgery
  Assessment of how patients perceive and feel about their physical appearance after the finalization of breast cancer treatments through the validated questionnaire Body Image Scale Questionnaire (BIS).

CONTACTS AND LOCATIONS:
Overall Officials: Berta Díaz-Feijoo, MD, PhD, Study Director — Hospital Clinic of Barcelona; Eduard Mension Coll, MD, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and ethical restrictions related to the confidentiality of patient information. The informed consent obtained from participants does not include provisions for data sharing beyond the primary research team.

REFERENCES:
- [Background] Angelats L, Pare L, Rubio-Perez C, Sanfeliu E, Gonzalez A, Segui E, Villacampa G, Marin-Aguilera M, Pernas S, Conte B, Albarran-Fernandez V, Martinez-Saez O, Aguirre A, Galvan P, Fernandez-Martinez A, Cobo S, Rey M, Martinez-Romero A, Walbaum B, Schettini F, Vidal M, Buckingham W, Munoz M, Adamo B, Agrawal Y, Guedan S, Pascual T, Agudo J, Grzelak M, Borcherding N, Heyn H, Vivancos A, Parker JS, Villagrasa P, Perou CM, Prat A, Braso-Maristany F. Linking tumor immune infiltration to enhanced longevity in recurrence-free breast cancer. ESMO Open. 2025 Jan;10(1):104109. doi: 10.1016/j.esmoop.2024.104109. Epub 2025 Jan 6. PMID 39765189
- [Background] Toohey K, Hunter M, McKinnon K, Casey T, Turner M, Taylor S, Paterson C. A systematic review of multimodal prehabilitation in breast cancer. Breast Cancer Res Treat. 2023 Jan;197(1):1-37. doi: 10.1007/s10549-022-06759-1. Epub 2022 Oct 21. PMID 36269525
- [Background] Denkert C, von Minckwitz G, Darb-Esfahani S, Lederer B, Heppner BI, Weber KE, Budczies J, Huober J, Klauschen F, Furlanetto J, Schmitt WD, Blohmer JU, Karn T, Pfitzner BM, Kummel S, Engels K, Schneeweiss A, Hartmann A, Noske A, Fasching PA, Jackisch C, van Mackelenbergh M, Sinn P, Schem C, Hanusch C, Untch M, Loibl S. Tumour-infiltrating lymphocytes and prognosis in different subtypes of breast cancer: a pooled analysis of 3771 patients treated with neoadjuvant therapy. Lancet Oncol. 2018 Jan;19(1):40-50. doi: 10.1016/S1470-2045(17)30904-X. Epub 2017 Dec 7. PMID 29233559
- [Background] Valenza C, Taurelli Salimbeni B, Santoro C, Trapani D, Antonarelli G, Curigliano G. Tumor Infiltrating Lymphocytes across Breast Cancer Subtypes: Current Issues for Biomarker Assessment. Cancers (Basel). 2023 Jan 26;15(3):767. doi: 10.3390/cancers15030767. PMID 36765724
- [Background] Wiggins JM, Opoku-Acheampong AB, Baumfalk DR, Siemann DW, Behnke BJ. Exercise and the Tumor Microenvironment: Potential Therapeutic Implications. Exerc Sport Sci Rev. 2018 Jan;46(1):56-64. doi: 10.1249/JES.0000000000000137. PMID 29166299
- [Background] van Waart H, Stuiver MM, van Harten WH, Geleijn E, Kieffer JM, Buffart LM, de Maaker-Berkhof M, Boven E, Schrama J, Geenen MM, Meerum Terwogt JM, van Bochove A, Lustig V, van den Heiligenberg SM, Smorenburg CH, Hellendoorn-van Vreeswijk JA, Sonke GS, Aaronson NK. Effect of Low-Intensity Physical Activity and Moderate- to High-Intensity Physical Exercise During Adjuvant Chemotherapy on Physical Fitness, Fatigue, and Chemotherapy Completion Rates: Results of the PACES Randomized Clinical Trial. J Clin Oncol. 2015 Jun 10;33(17):1918-27. doi: 10.1200/JCO.2014.59.1081. Epub 2015 Apr 27. PMID 25918291
- [Background] Cannioto RA, Hutson A, Dighe S, McCann W, McCann SE, Zirpoli GR, Barlow W, Kelly KM, DeNysschen CA, Hershman DL, Unger JM, Moore HCF, Stewart JA, Isaacs C, Hobday TJ, Salim M, Hortobagyi GN, Gralow JR, Albain KS, Budd GT, Ambrosone CB. Physical Activity Before, During, and After Chemotherapy for High-Risk Breast Cancer: Relationships With Survival. J Natl Cancer Inst. 2021 Jan 4;113(1):54-63. doi: 10.1093/jnci/djaa046. PMID 32239145
- [Background] Peterson LL, Ligibel JA. Physical Activity and Breast Cancer: an Opportunity to Improve Outcomes. Curr Oncol Rep. 2018 Apr 30;20(7):50. doi: 10.1007/s11912-018-0702-1. PMID 29713835
- [Background] Ochoa-Arnedo C, Prats C, Travier N, Marques-Feixa L, Flix-Valle A, de Frutos ML, Domingo-Gil E, Medina JC, Serra-Blasco M. Stressful Life Events and Distress in Breast Cancer: A 5-Years Follow-Up. Int J Clin Health Psychol. 2022 May-Aug;22(2):100303. doi: 10.1016/j.ijchp.2022.100303. Epub 2022 Apr 1. PMID 35572072
- [Background] Oh PJ, Shin SR, Ahn HS, Kim HJ. Meta-analysis of psychosocial interventions on survival time in patients with cancer. Psychol Health. 2016;31(4):396-419. doi: 10.1080/08870446.2015.1111370. Epub 2015 Dec 18. PMID 26518363
- [Background] Andersen BL, Yang HC, Farrar WB, Golden-Kreutz DM, Emery CF, Thornton LM, Young DC, Carson WE 3rd. Psychologic intervention improves survival for breast cancer patients: a randomized clinical trial. Cancer. 2008 Dec 15;113(12):3450-8. doi: 10.1002/cncr.23969. PMID 19016270
- [Background] Chen Y, Ahmad M. Effectiveness of adjunct psychotherapy for cancer treatment: a review. Future Oncol. 2018 Jun;14(15):1487-1496. doi: 10.2217/fon-2017-0671. Epub 2018 May 16. PMID 29767550
- [Background] Tommasi C, Balsano R, Coriano M, Pellegrino B, Saba G, Bardanzellu F, Denaro N, Ramundo M, Toma I, Fusaro A, Martella S, Aiello MM, Scartozzi M, Musolino A, Solinas C. Long-Term Effects of Breast Cancer Therapy and Care: Calm after the Storm? J Clin Med. 2022 Dec 6;11(23):7239. doi: 10.3390/jcm11237239. PMID 36498813
- [Background] Santa Mina D, Brahmbhatt P, Lopez C, Baima J, Gillis C, Trachtenberg L, Silver JK. The Case for Prehabilitation Prior to Breast Cancer Treatment. PM R. 2017 Sep;9(9S2):S305-S316. doi: 10.1016/j.pmrj.2017.08.402. PMID 28942905
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Long-term outcomes for neoadjuvant versus adjuvant chemotherapy in early breast cancer: meta-analysis of individual patient data from ten randomised trials. Lancet Oncol. 2018 Jan;19(1):27-39. doi: 10.1016/S1470-2045(17)30777-5. Epub 2017 Dec 11. PMID 29242041
- See also: Breast cancer statistics — http://www.cancer.net/cancer-types/breast-cancer/statistics